CLINICAL TRIAL: NCT04985591
Title: The Effect of Liposuction on Menses: a Retrospective Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH9H-2019-T221-2
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Menstrual Irregularity
MeSH Terms: conditions — Menstruation Disturbances | interventions — Lipectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liposuction group (Experimental)
  Interventions: Procedure: Liposuction
- Other plastic surgery group (Placebo Comparator)
  Interventions: Procedure: Other plastic surgery

INTERVENTIONS:
Procedure: Liposuction — A small, inconspicuous incision was made in the liposuction group to dislodge fat out of the body.
  Arms: liposuction group
Procedure: Other plastic surgery — Other plastic surgery like blepharoplasty or keloid excision.
  Arms: Other plastic surgery group

SUMMARY:
The prevalence of obesity nearly tripled from 1975 to 2021, resulting in liposuction, as an effective shaping method, to be performed more frequently. Liposuction is a surgical procedure that uses a specialized instrument to suck fat fragments in the subcutaneous fat layer through a small incision. Analyzing a large sample sizes of patients who had liposuction, we found that some female patients underwent menstrual irregularity after liposuction. In 2004, Carolyn et al. reported several cases in which there was a connection between liposuction and an early onset of menses. Further studies showed that an early onset of menses may be related to the volume of adipose tissue extracted, the amount of anesthesia given, the area of liposuction, and body weight. However, the sample of that study was small, as there were only 17 cases included in the statistical model, and there are few articles in which the impact of liposuction on menses has been studied. To better understand whether menstrual irregularity will occur after liposuction, patients with postmenopausal or preoperative menstrual irregularity were excluded, leaving a sample of 518 female patients to be reviewed. A better understanding of the impact of liposuction on menses may help clinical doctors predict the underlying risk of menstrual irregularity after liposuction and identify individuals at higher risk. The findings may contribute to further understanding of menstrual irregularity.

ELIGIBILITY:
Inclusion Criteria:patients who were in 18-55 and have a regular menses -

Exclusion Criteria:Patients who were younger than 18 years old or older than 55 years old, who were in the perimenopausal or postmenopausal stage or who had menstrual irregularity before plastic surgery were excluded from both groups.

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 516 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
menstrual irregularity | three months
  to detect any change in the menses during the following 3 months, post surgery

IPD SHARING:
Plan to Share IPD: No